CLINICAL TRIAL: NCT00048100
Title: Anti-Leukemic Dendritic Cell Activated Donor Lymphocytes for Therapy of Relapsed Leukemia After Allogeneic Stem Cell Therapy
Brief Title: Anti-Leukemic Dendritic Cell Activated Donor Lymphocytes
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Slow accrual.
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ID00-034
Record Dates: First submitted 2002-10-24; First posted 2002-10-25 (Estimated); Last update posted 2018-10-31 (Actual); Status verified 2018-10

CONDITIONS: Leukemia, Myelocytic, Acute
Keywords: Dendritic cells; Lymphocytes; AML
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Blood Component Removal; Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Apheresis + Transplant (Experimental): Skin biopsy & either a leukodepletion apheresis or an additional marrow aspiration prior to marrow or stem cell transplantation.
  Interventions: Procedure: Apheresis; Biological: Stem Cell Transplant

INTERVENTIONS:
Procedure: Apheresis — Apheresis for T-Cell collection
Biological: Stem Cell Transplant — Stem cell or marrow infusions of allogeneic donor lymphocytes activated by acute leukemia derived dendritic cells (DC/ADL).
  Other Names: SCT; Stem Cell Transplantation

SUMMARY:
Objectives:

1. Determine the toxicity of infusions of allogeneic donor lymphocytes activated by acute leukemia derived dendritic cells (DC/ADL) in relapsed patients after allo-stem cell transplants.
2. Quantitate the alloreactivity of DC/ADL and circulating immune effector cells in patients after infusion.
3. Assess efficacy of acute myelogenous leukemia (AML) or Chronic Myelogenous Leukemia in Blastic Crisis (CML-BC) derived dendritic cells and activated lymphocytes in promoting and sustaining remission in patients with relapse after allo-BMT or stem cell transplant.

ELIGIBILITY:
Inclusion Criteria:

* AML (any type except M3) or CIVIL in blast crisis with greater than or equal to 20% bone marrow blasts at the time of related donor marrow or stem cell transplantation or at relapse post transplant.
* Willing to undergo a skin biopsy and either a leukodepletion apheresis or an additional marrow aspiration.
* Stem cell or marrow donor willing to have apheresis for T-Cell collection.
* Written voluntary informed consent must be obtained from patient and donor.

Exclusion Criteria:

* Medical, social or psychologic factors which would prevent the patient from receiving or cooperating with the full course of therapy or understanding the informed consent procedure.
* AML French-American-British (FAB) subtype M3.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2001-02; Primary Completion 2005-05 (Actual); Study Completion 2005-05 (Actual)

PRIMARY OUTCOMES:
Participant Toxicity Levels | From stem cell transplant baseline to 30 plus days post transplant.
  Participant toxicity of infusions of allogeneic donor lymphocytes activated by acute leukemia derived dendritic cells (DC/ADL) in relapsed patients after allo-stem cell transplants.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth J. Shpall, MD, Principal Investigator — UT MD Anderson Cancer Center
Locations (1):
- M.D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center website — http://www.mdanderson.org